CLINICAL TRIAL: NCT00590070
Title: Randomized Evaluation Of Intracoronary Nitroprusside vs Adenosine After Thrombus-aspiration During Primary PErcutaneous Coronary Intervention for the Prevention of No Reflow in Acute Myocardial Infarction
Brief Title: THE REOPEN-AMI STUDY - Intracoronary Nitroprusside Versus Adenosine in Acute Myocardial Infarction
Acronym: REOPEN-AMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, GIANPAOLO NICCOLI, Dott. Prof., Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REOPEN-AMI 2007-006794-93; 2007-006794-93
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; no reflow; primary PCI; Coronary no-reflow phenomenon; primary percutaneous coronary intervention (primary PCI)
MeSH Terms: conditions — Myocardial Infarction | interventions — Adenosine; Nitroprusside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Patients will receive intravenous administration of abciximab prior to PCI. After wire crossing, thrombus aspiration will be performed. The device will removed outside the body, flushed with saline and subsequently reintroduced in the culprit vessel beyond the occlusion site and intracoronary drugs will be selectively administered.
  Interventions: Drug: adenosine
- 2 (Active Comparator): Patients will receive intravenous administration of abciximab prior to PCI. After wire crossing, thrombus aspiration will be performed. The device will removed outside the body, flushed with saline and subsequently reintroduced in the culprit vessel beyond the occlusion site and intracoronary drugs will be selectively administered.
  Interventions: Drug: nitroprusside
- 3 (Placebo Comparator): Patients will receive intravenous administration of abciximab prior to PCI. After wire crossing, thrombus aspiration will be performed. The device will removed outside the body, flushed with saline and subsequently reintroduced in the culprit vessel beyond the occlusion site and intracoronary drugs will be selectively administered
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: adenosine — Adenosine (80 mcg as fast bolus followed by 2 mg given in 33cc of saline in 2 minutes as slow bolus)
  Arms: 1
Drug: nitroprusside — Nitroprusside (60 mcg as fast bolus followed by 100 mcg given in 33cc of 5% glucose in 2 minutes as slow bolus)
  Arms: 2
Drug: placebo — 33 cc of heparinized saline given in 2 minutes as slow bolus
  Arms: 3

SUMMARY:
The occurrence of no-reflow phenomenon after recanalization of the infarct related artery in acute myocardial infarction is described in up to 40% of cases. This event is associated with a worse prognosis at follow up and an unfavourable left ventricular remodelling . Two main pathogenetic mechanisms cause no-reflow: distal embolization and ischemia-reperfusion injury.

Due to the multifactorial pathogenesis of no-reflow during acute MI a combined mechanic and pharmacologic approach is believed to offer a better solution for achieving optimal microvascular reperfusion. Thus, in this randomized study we will assess the effect of nitroprusside or adenosine in adjunct to current best therapy (thrombus aspiration and IIb-IIIa antagonists) for ST elevation MI using ST segment resolution on standard 12 leads ECG as primary endpoint of myocardial reperfusion.

DETAILED DESCRIPTION:
The occurrence of no-reflow phenomenon after recanalization of the infarct related artery in acute myocardial infarction is described in up to 40% of cases. This event is associated with a worse prognosis at follow up and an unfavourable left ventricular remodelling. Two main pathogenetic mechanisms cause no-reflow: distal embolization and ischemia-reperfusion injury. Microembolization, which may be well prevented by a mechanic approach (device-based), play of course an important role in the no-reflow during primary percutaneous coronary intervention (primary PCI), however ischemia reperfusion injury is also independent of microemboli, indeed it occurs in the animal model after ligation of a non atherosclerotic coronary. Thrombus aspiration assisted primary intervention achieves complete resolution of the ST segment in 60% only of patients, whereas results of filter based studies have been substantially negative. A recent meta-analysis confirmed that thrombus aspiration improves microvascular perfusion, whereas filters do not.

Taken together available data suggest that other approach need to be tested in conjunction with the mechanical one to further improve microvascular integrity in this setting. Importantly, current antiplatelet therapy during reperfusion therapy for acute MI has not abolished the no-reflow phenomenon. Based on the experience matured in many studies of basic cardiology which investigated the model of ischemia and reperfusion various drugs have been tested in the human model.

Two drugs have emerged in particular as possible adjunct to reperfusion therapy: nitroprusside and adenosine. For the former good results have been obtained in small series, in contrast adenosine has been tested in a large randomized trial (AMISTAD-II trial) with controversial results when used at low dose. Another study using larger doses and a sub-analysis of a high dose group of the AMISTAD-II trial suggested a beneficial effect on infarct size. Importantly, none of this studies have been performed in the setting of thrombus aspiration.

Due to the multifactorial pathogenesis of no-reflow during acute MI a combined mechanic and pharmacologic approach is believed to offer a better solution for achieving optimal microvascular reperfusion. Thus, in this randomized study we will assess the effect of nitroprusside or adenosine in adjunct to current best therapy (thrombus aspiration and IIb-IIIa antagonists) for ST elevation MI using ST segment resolution on standard 12 leads ECG as primary endpoint of myocardial reperfusion.

Study Design

The REOPEN-AMI will be a placebo-controlled, randomized, open label, blind-examination (PROBE), multicenter, trial of the effects of intracoronary adenosine or nitroprusside on coronary reflow in patients undergoing primary or rescue PCI and thrombus-aspiration. The recruiting period comprises 1 year time between January 2008 and December 2008. During the last months, the others participating centres in Italy, were contacted and entered in the study after agreement. As result prospective recruitment should start at the same time in all participating centers. Each center, to be activated for the study, had to warrant (fully describing the search process as well as the characteristics of the internal database) ability to provide detailed data regarding all the patients.

The study protocol complied with the declaration of Helsinki and has been approved by the ethics committee of the coordinating center. Informed consent to both the treated group ( adenosine or nitroprusside) or placebo will have to be obtained for each patient enrolled in the study

METHODS

All patient will receive intravenous administration of abciximab prior to PCI. After wire crossing, thrombus aspiration will be performed. The device will removed outside the body, flushed with saline and subsequently reintroduced in the culprit vessel beyond the occlusion site and intracoronary drugs will be selectively administered. At this stage the patient will be randomized either to intracoronary Adenosine (80 mcg as fast bolus followed by 2 mg given in 33cc of saline in 2 minutes as slow bolus), nitroprusside (60 mcg as fast bolus followed by 100 mcg given in 33cc of 5% glucose in 2 minutes as slow bolus) or placebo (33 cc of heparinized saline given in 2 minutes as slow bolus). Due to the short half-life of both drugs we have chosen a bolus plus infusion regimen in order to allow a more sustained effect of the two drugs on the microcirculation. The safety and efficacy of this drug regimen has been tested in a small pilot study in our catheterization laboratory. We have compared the two drugs regimens to traditional single bolus administration of adenosine for the evaluation of fractional flow reserve (FFR) in ten patients (5 for adenosine and 5 for nitroprusside) undergoing pressure wire evaluation of an intermediate stenosis. We found similar FFR in both groups but more prolonged dilatation of the microcirculation compared to group of traditional single bolus adenosine administration (data not shown).

If the thrombus aspiration device cannot be advanced for mechanical reasons in the culprit vessel, drugs administration will be performed trough the guiding catheter after predilatation. Data will be analyzed according to the intention to treat principle.

Angiographic measures

Coronary angiograms will be obtained with the aim of facilitating angiographic analyses (long acquisition without magnification). All CDs of primary PCI will be sent to the coordinator center where they will be processed by extrapolating the images regarding baseline, thrombus aspiration, diver reintroduction in the culprit lesion beyond the occlusion site and the post-PCI view. The core laboratory for centralized, blind analyses will be the Catholic University of Rome. For each patient coronary angiograms will be analyzed to assess the following:

* Antegrade coronary flow according to the standard TIMI criteria flow
* Corrected TIMI Frame Count according to Gibson
* MBG according to van't Hof et al.
* Thrombus score according to TIMI study group (0= no cineangiographic characteristics of thrombus are present; 1 = possible thrombus is present with such angiography characteristics as reduced contrast density, haziness, irregular lesion contour, or a smooth convex meniscus at the site of total occlusion suggestive but not diagnostic of thrombus. 2 = definite thrombus, with greatest dimension <1/2 the vessel diameter; 3 = definite thrombus , with greatest linear dimension >1/2 but <2 vessel diameters; 4 = definite thrombus, with the largest dimension >2 vessel diameters ; 5= there is a total occlusion);
* collateral grade according to Rentrop Angiographic "no-reflow" will be defined as a final TIMI flow ≤ 2 or TIMI flow 3 with a MBG < 2.

Intracoronary ECG

Monitoring of intracoronary ST segment during PCI, up to the end of the procedure will be performed according to flow chart . The technique has been described elsewhere (22). Briefly, the proximal end of the wire chosen for recanalization will be used as a unipolar derivation which substitutes the V5 leads on precordial ECG. ST resolution will be monitored during the procedure and ECG acquisition will be done at baseline, after effective thrombus aspiration, after intracoronary drugs administration and at the end of the procedure. Each ECG will be quantitatively assessed. Lack of resolution will be defined as a ST elevation resolution of < 30%. Partial resolution will be considered a ST resolution ≥30% but <70%. Furthermore times needed to obtain full or partial ST resolution will be recorded. Anginal pain at starting and at each time points will be assessed.

12-leads surface ECG After the procedure, at 90 min, a standard 12 leads ECG will be used for evaluating ST resolution both on single lead, showing maximal ST elevation, and on the sum of multiple leads, showing ST elevation on admission. Lack of ST resolution will be defined as an ST resolution <30%. Partial resolution as an ST resolution <70% but > 30%. The detailed analysis of ECG resolution has been described elsewhere. The core laboratory for intracoronary or surface ECG analysis will be the Catholic University of Rome.

Contrast and bidimensional echocardiography

Echocontrastographic evaluation of reperfusion will be carried out on day 7. Echocontrastographic definition of no reflow is, according to previously described methods, when > 25% of dysfunctioning segments had reduced or absent opacification (score 2-3). The technique has been described elsewhere. Briefly, myocardial contrast echocardiography studies will be performed using real-time contrast pulse sequencing operating on a Sequoia ultrasound system (Siemens, Malvern, Pennsylvania). Contrast pulse sequencing is a novel real-time MCE method that, thanks to the analysis of non-linear response of contrast bubbles in fundamental and higher harmonics, is able to provide an image with excellent signal-to-noise ratio and with particularly high sensitivity and penetration using a very low mechanical index. A second-generation ultrasound contrast agent Sonovue (Bracco, Milan, Italy) will be administered intravenously (5 ml at 1 ml/min). Myocardial opacification at MCE will be visually assessed in each of the 16 myocardial segments and semiquantitatively scored. Single perfusion score will be assigned on the basis of both the change in myocardial signal intensity throughout the replenishment curve and the degree of opacification at the peak contrast effect. Scores were graded as 1 = normal, 2 = reduced, or 3 = absent opacification. A contrast score index (CSI) will be calculated by the sum of MCE score in each segment divided by the total number of segments..

Echocardiographic evaluation will be obtained on day 7 and at follow up (6 months). Regional wall motion (WM) will be semiquantitatively scored by 2 experienced blinded observers according to the recommendations of the American Society of Echocardiography (1 = normal, 2 = hypokinesia, 3 = akinesia, 4 = dyskinesia) and a wall motion score index (WMSI) will be calculated by the sum of the score of all segments divided by the total number of segments. Left ventricular (LV) volumes will be calculated by the modified Simpson biplane method. Endocardial length of severe WM abnormality (WM score = 3) (WML) and of transmural contrast defect (CD score = 3) (CDL) will be calculated in each apical view, averaged, and expressed as a percentage of LV length.

Ejection fraction will be calculated from the formula: (end-diastolic volume end-systolic volume)/end diastolic volume. Functional improvement at 6 months will be calculated as percentage change of WMSI at 6 months compared to 7 day. Temporal changes in LV volumes will be calculated as the percentage changes at 6 months compared to baseline. Left ventricular remodelling will be considered as an increase in LV end-diastolic volume > 20% at 6 months compared to baseline (25-26). The core laboratory for the echocardiographic analysis will be the Catholic University of Rome.

Clinical follow-up

The incidence of cardiac death, myocardial infarction, target lesion revascularization and heart failure requiring hospitalization will be assessed at 6 months and 1 year by telephone contact. A cumulative of such end-points will be defined as major adverse cardiac events (MACEs).

Endpoints of the study

Primary end-point of the study will be rate of ST resolution on surface ECG. Secondary end-points will be: 1) rate of angiographic no-reflow; 2) changes of LV volumes at follow-up; 3) rate of no-reflow on IC ECG; 4) rate of no-reflow at echocontrastography; 5) rate of MACEs.

Statistical analysis and sample size calculation Data distribution will be assessed by the Kolgomorov-Smirnov test. Comparison between groups will be performed by Anova or Kruskall-Wallis test as appropriate. Post-hoc comparison will be performed with the Bonferroni correction. Comparison between categorical variable will be done using the Fischer exact test. Student T test for dependent variables will be used to compare changes in LV volumes in each group over time and interaction assessed by Anova. Pre-specified sub-group analysis according to main clinical and angiographic data will be also performed, in order to identify subgroups of patients who may have a particular benefit from treatments.

Sample size is calculated as follow. Considering an effect size of 0.2 (improvement of the primary endpoint by 20%, which is obtained considering an ST resolution of 50% in the placebo group and an ST resolution of 70% in the treatment groups), a power of 0.8 and an alfa of 0.05, with 2 degree of freedom the required sample size is 240 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms onset < 12 hours prior to enrollment
2. ST-segment elevation of at least 2 mm in two or more contiguous leads
3. TIMI flow 0-1 at baseline angiography

Exclusion Criteria:

Demographic, history and clinical examination

1. age less than 18 years
2. previous STEMI
3. patients presenting in cardiogenic shock
4. pregnancy
5. patients with renal failure
6. contraindications to contrast agents, which cannot be managed medically or study medications, including aspirin, clopidogrel and ticlopidine, and heparin

   Electrocardiogram
7. left bundle branch block, paced rhythm, frequent ventricular ectopy, pre-excitation or other conditions or artifacts interfering with interpretation of ST segment resolution Angiography
8. culprit lesion located in a by-pass graft
9. stent thrombosis
10. culprit lesion non identified
11. left main disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Rate of major adverse cardiac events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Niccoli, MD, PhD, Principal Investigator — Institute of Cardiology UCSC; Filippo Crea, MD, Study Chair — Institute of Cardiology UCSC
Locations (1):
- Dipartimento Medicina Cardiovascolare, Rome, Rome, Italy

REFERENCES:
- [Background] Ito H, Okamura A, Iwakura K, Masuyama T, Hori M, Takiuchi S, Negoro S, Nakatsuchi Y, Taniyama Y, Higashino Y, Fujii K, Minamino T. Myocardial perfusion patterns related to thrombolysis in myocardial infarction perfusion grades after coronary angioplasty in patients with acute anterior wall myocardial infarction. Circulation. 1996 Jun 1;93(11):1993-9. doi: 10.1161/01.cir.93.11.1993. PMID 8640973
- [Background] Ito H, Tomooka T, Sakai N, Yu H, Higashino Y, Fujii K, Masuyama T, Kitabatake A, Minamino T. Lack of myocardial perfusion immediately after successful thrombolysis. A predictor of poor recovery of left ventricular function in anterior myocardial infarction. Circulation. 1992 May;85(5):1699-705. doi: 10.1161/01.cir.85.5.1699. PMID 1572028
- [Background] Rezkalla SH, Kloner RA. No-reflow phenomenon. Circulation. 2002 Feb 5;105(5):656-62. doi: 10.1161/hc0502.102867. No abstract available. PMID 11827935
- [Background] Henriques JP, Zijlstra F, Ottervanger JP, de Boer MJ, van 't Hof AW, Hoorntje JC, Suryapranata H. Incidence and clinical significance of distal embolization during primary angioplasty for acute myocardial infarction. Eur Heart J. 2002 Jul;23(14):1112-7. doi: 10.1053/euhj.2001.3035. PMID 12090749
- [Background] Reffelmann T, Kloner RA. The no-reflow phenomenon: A basic mechanism of myocardial ischemia and reperfusion. Basic Res Cardiol. 2006 Sep;101(5):359-72. doi: 10.1007/s00395-006-0615-2. PMID 16915531
- [Background] Burzotta F, Trani C, Romagnoli E, Mazzari MA, Rebuzzi AG, De Vita M, Garramone B, Giannico F, Niccoli G, Biondi-Zoccai GG, Schiavoni G, Mongiardo R, Crea F. Manual thrombus-aspiration improves myocardial reperfusion: the randomized evaluation of the effect of mechanical reduction of distal embolization by thrombus-aspiration in primary and rescue angioplasty (REMEDIA) trial. J Am Coll Cardiol. 2005 Jul 19;46(2):371-6. doi: 10.1016/j.jacc.2005.04.057. PMID 16022970
- [Background] Stone GW, Webb J, Cox DA, Brodie BR, Qureshi M, Kalynych A, Turco M, Schultheiss HP, Dulas D, Rutherford BD, Antoniucci D, Krucoff MW, Gibbons RJ, Jones D, Lansky AJ, Mehran R; Enhanced Myocardial Efficacy and Recovery by Aspiration of Liberated Debris (EMERALD) Investigators. Distal microcirculatory protection during percutaneous coronary intervention in acute ST-segment elevation myocardial infarction: a randomized controlled trial. JAMA. 2005 Mar 2;293(9):1063-72. doi: 10.1001/jama.293.9.1063. PMID 15741528
- [Background] Cura FA, Escudero AG, Berrocal D, Mendiz O, Trivi MS, Fernandez J, Palacios A, Albertal M, Piraino R, Riccitelli MA, Gruberg L, Ballarino M, Milei J, Baeza R, Thierer J, Grinfeld L, Krucoff M, O'Neill W, Belardi J; PREMIAR Investigators. Protection of Distal Embolization in High-Risk Patients with Acute ST-Segment Elevation Myocardial Infarction (PREMIAR). Am J Cardiol. 2007 Feb 1;99(3):357-63. doi: 10.1016/j.amjcard.2006.08.038. Epub 2006 Dec 13. PMID 17261398
- [Background] Burzotta F, Testa L, Giannico F, Biondi-Zoccai GG, Trani C, Romagnoli E, Mazzari M, Mongiardo R, Siviglia M, Niccoli G, De Vita M, Porto I, Schiavoni G, Crea F. Adjunctive devices in primary or rescue PCI: a meta-analysis of randomized trials. Int J Cardiol. 2008 Jan 24;123(3):313-21. doi: 10.1016/j.ijcard.2006.12.018. Epub 2007 Mar 26. PMID 17383756
- [Background] Chaitman BR, Lim MJ. No reflow and the quest to achieve optimal perfusion during the acute phase of myocardial infarction. J Am Coll Cardiol. 2004 Jul 21;44(2):313-5. doi: 10.1016/j.jacc.2004.04.020. No abstract available. PMID 15261924
- [Background] Hillegass WB, Dean NA, Liao L, Rhinehart RG, Myers PR. Treatment of no-reflow and impaired flow with the nitric oxide donor nitroprusside following percutaneous coronary interventions: initial human clinical experience. J Am Coll Cardiol. 2001 Apr;37(5):1335-43. doi: 10.1016/s0735-1097(01)01138-x. PMID 11300444
- [Background] Marzilli M, Orsini E, Marraccini P, Testa R. Beneficial effects of intracoronary adenosine as an adjunct to primary angioplasty in acute myocardial infarction. Circulation. 2000 May 9;101(18):2154-9. doi: 10.1161/01.cir.101.18.2154. PMID 10801755
- [Background] Ota S, Nishikawa H, Takeuchi M, Nakajima K, Nakamura T, Okamoto S, Setsuda M, Makino K, Yamakado T, Nakano T. Impact of nicorandil to prevent reperfusion injury in patients with acute myocardial infarction: Sigmart Multicenter Angioplasty Revascularization Trial (SMART). Circ J. 2006 Sep;70(9):1099-104. doi: 10.1253/circj.70.1099. PMID 16936418
- [Background] Amit G, Cafri C, Yaroslavtsev S, Fuchs S, Paltiel O, Abu-Ful A, Weinstein JM, Wolak A, Ilia R, Zahger D. Intracoronary nitroprusside for the prevention of the no-reflow phenomenon after primary percutaneous coronary intervention in acute myocardial infarction. A randomized, double-blind, placebo-controlled clinical trial. Am Heart J. 2006 Nov;152(5):887.e9-14. doi: 10.1016/j.ahj.2006.05.010. PMID 17070151
- [Background] Pasceri V, Pristipino C, Pelliccia F, Granatelli A, Speciale G, Roncella A, Pironi B, Capasso M, Richichi G. Effects of the nitric oxide donor nitroprusside on no-reflow phenomenon during coronary interventions for acute myocardial infarction. Am J Cardiol. 2005 Jun 1;95(11):1358-61. doi: 10.1016/j.amjcard.2005.01.082. PMID 15904643
- [Background] Ross AM, Gibbons RJ, Stone GW, Kloner RA, Alexander RW; AMISTAD-II Investigators. A randomized, double-blinded, placebo-controlled multicenter trial of adenosine as an adjunct to reperfusion in the treatment of acute myocardial infarction (AMISTAD-II). J Am Coll Cardiol. 2005 Jun 7;45(11):1775-80. doi: 10.1016/j.jacc.2005.02.061. PMID 15936605
- [Background] TIMI Study Group. The Thrombolysis in Myocardial Infarction (TIMI) trial. Phase I findings. N Engl J Med. 1985 Apr 4;312(14):932-6. doi: 10.1056/NEJM198504043121437. No abstract available. PMID 4038784
- [Background] Gibson CM, Cannon CP, Daley WL, Dodge JT Jr, Alexander B Jr, Marble SJ, McCabe CH, Raymond L, Fortin T, Poole WK, Braunwald E. TIMI frame count: a quantitative method of assessing coronary artery flow. Circulation. 1996 Mar 1;93(5):879-88. doi: 10.1161/01.cir.93.5.879. PMID 8598078
- [Background] Gibson CM, de Lemos JA, Murphy SA, Marble SJ, McCabe CH, Cannon CP, Antman EM, Braunwald E; TIMI Study Group. Combination therapy with abciximab reduces angiographically evident thrombus in acute myocardial infarction: a TIMI 14 substudy. Circulation. 2001 May 29;103(21):2550-4. doi: 10.1161/01.cir.103.21.2550. PMID 11382722
- [Background] Rentrop KP, Cohen M, Blanke H, Phillips RA. Changes in collateral channel filling immediately after controlled coronary artery occlusion by an angioplasty balloon in human subjects. J Am Coll Cardiol. 1985 Mar;5(3):587-92. doi: 10.1016/s0735-1097(85)80380-6. PMID 3156171
- [Background] Friedman PL, Shook TL, Kirshenbaum JM, Selwyn AP, Ganz P. Value of the intracoronary electrocardiogram to monitor myocardial ischemia during percutaneous transluminal coronary angioplasty. Circulation. 1986 Aug;74(2):330-9. doi: 10.1161/01.cir.74.2.330. PMID 2942314
- [Background] Schroder R, Dissmann R, Bruggemann T, Wegscheider K, Linderer T, Tebbe U, Neuhaus KL. Extent of early ST segment elevation resolution: a simple but strong predictor of outcome in patients with acute myocardial infarction. J Am Coll Cardiol. 1994 Aug;24(2):384-91. doi: 10.1016/0735-1097(94)90292-5. PMID 8034872
- [Background] Galiuto L, Garramone B, Burzotta F, Lombardo A, Barchetta S, Rebuzzi AG, Crea F; REMEDIA Investigators. Thrombus aspiration reduces microvascular obstruction after primary coronary intervention: a myocardial contrast echocardiography substudy of the REMEDIA Trial. J Am Coll Cardiol. 2006 Oct 3;48(7):1355-60. doi: 10.1016/j.jacc.2006.05.059. Epub 2006 Sep 14. PMID 17010794
- [Background] Bolognese L, Carrabba N, Parodi G, Santoro GM, Buonamici P, Cerisano G, Antoniucci D. Impact of microvascular dysfunction on left ventricular remodeling and long-term clinical outcome after primary coronary angioplasty for acute myocardial infarction. Circulation. 2004 Mar 9;109(9):1121-6. doi: 10.1161/01.CIR.0000118496.44135.A7. Epub 2004 Feb 16. PMID 14967718
- [Background] Bolognese L, Cerisano G, Buonamici P, Santini A, Santoro GM, Antoniucci D, Fazzini PF. Influence of infarct-zone viability on left ventricular remodeling after acute myocardial infarction. Circulation. 1997 Nov 18;96(10):3353-9. doi: 10.1161/01.cir.96.10.3353. PMID 9396427